CLINICAL TRIAL: NCT02502760
Title: Using Multimodal Prehabilitation to Improve Outcomes for Frail Patients Undergoing Resection of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Franco Carli, Professor, Montreal General Hospital Department of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-131-MUHC
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Neoplasms
Keywords: Postoperative Complications; Perioperative Care; Colorectal Surgery; Frail Elderly
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): Immediately after randomization and until surgery, patients in this arm will:
  1. - Receive a personalized physical exercise program
  2. - Receive nutritional counselling with Whey protein isolate powder
  3. - Receive relaxation techniques
  Interventions: Behavioral: Physical Exercise Program; Dietary Supplement: Whey Protein Isolate Powder; Behavioral: Relaxation Techniques
- Rehabilitation (Active Comparator): Patients in this arm will receive the same personalized physical exercise program, nutritional intervention and relaxation techniques as patients in the other arm but to be started after surgery.
  Interventions: Behavioral: Physical Exercise Program; Dietary Supplement: Whey Protein Isolate Powder; Behavioral: Relaxation Techniques

INTERVENTIONS:
Behavioral: Physical Exercise Program — Physical exercises personalized by a kinesiologist consisting of walking or stationary bike and elastic band exercises.
Dietary Supplement: Whey Protein Isolate Powder — Nutritional counselling is given to patients to ensure their daily proteins and energy requirements are met. Whey Protein Isolate Powder (Immunocal) is provided.
  Immunocal1.5g/kg PO (by mouth) per day separated in 2 daily doses
Behavioral: Relaxation Techniques — Relaxation techniques consisting of breathing exercises and using a relaxation CD.

SUMMARY:
The purpose of this study is to determine if a program of physical activity, nutritional supplements and relaxation techniques is effective at decreasing post operative complications in frail colorectal cancer patients undergoing resection.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patient undergoing resection
* Frail or intermediately frail patients (Fried score 2 and above)

Exclusion Criteria:

* Unable to communicate in French or English
* Premorbid conditions contraindicating physical exercise (dementia, Parkinson Disease, previous stroke with paresis, taking carbidopa/levodopa, donepezil or antidepressants)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08; Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Post operative complications | 30 days after surgery
  Comprehensive Complication Index (CCI)

SECONDARY OUTCOMES:
6 Minutes Walk Test Distance | 4 weeks after discharge
Hospital Length of Stay | 3-6 days
Readmission rates | 30 days after discharge
Anxiety and Depression | 30 days after discharge
  Using the Hospital Anxiety Depression Scale (HADS)
Health Related Quality of Life | 30 days after discharge
  Using the Short Form Health Survey (SF-36)

OTHER OUTCOMES:
Cost Effectiveness of treatment | 30 days after hospital discharge
  Factoring the cost of the program versus possible savings related to other primary and secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, MPhil, Principal Investigator — Professor, Department of Anesthesia
Locations (2):
- Canada (2):
  - McGill University Health Center; Montreal General Hospital, Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252
- [Derived] Carli F, Bousquet-Dion G, Awasthi R, Elsherbini N, Liberman S, Boutros M, Stein B, Charlebois P, Ghitulescu G, Morin N, Jagoe T, Scheede-Bergdahl C, Minnella EM, Fiore JF Jr. Effect of Multimodal Prehabilitation vs Postoperative Rehabilitation on 30-Day Postoperative Complications for Frail Patients Undergoing Resection of Colorectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Mar 1;155(3):233-242. doi: 10.1001/jamasurg.2019.5474. PMID 31968063